CLINICAL TRIAL: NCT00002100
Title: Phase I/II Study of Curdlan Sulfate
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AJI Pharma USA (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Purpose: Treatment
Other Study IDs: 127A; LCPL 92-1-28
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1994-04

CONDITIONS: HIV Infections
Keywords: Acquired Immunodeficiency Syndrome; AIDS-Related Complex; curdlan sulfate
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome; AIDS-Related Complex | interventions — curdlan sulfate

INTERVENTIONS:
Drug: Curdlan sulfate

SUMMARY:
To assess the safety and tolerance of curdlan sulfate, as well as its anti-HIV activity, in HIV-infected patients with CD4 T-lymphocytes less than 500 cells/mm3, using first single doses and then, after FDA review, daily doses for 7 days.

DETAILED DESCRIPTION:
In Phase I of the study, escalating single doses of intravenous curdlan sulfate are tested. In Phase II, curdlan sulfate is administered daily for 7 days. (NOTE: Phase I is completed.)

ELIGIBILITY:
Inclusion Criteria

Patients must have:

* HIV seropositivity.
* No current AIDS-defining opportunistic infection, lymphoma, Kaposi's sarcoma, or other malignancy.
* CD4 count < 500 cells/mm3.
* No critical illness that would shorten life expectancy to < 16 weeks.

Exclusion Criteria

Concurrent Medication:

Excluded:

* Antiretroviral or other experimental therapies.
* Anticoagulants.
* Steroids.
* Cytotoxic or immunosuppressive agents.

Concurrent Treatment:

Excluded:

* Radiotherapy.

Patients with the following prior condition are excluded:

History of heparin sensitivity.

Prior Medication:

Excluded within 1 month prior to study entry:

* Antiretroviral or other experimental therapies.
* Anticoagulants.
* Steroids.
* Cytotoxic or immunosuppressive agents.

Prior Treatment:

Excluded:

* Radiotherapy within 1 month prior to study entry. Active IV drug abuse.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult

CONTACTS AND LOCATIONS:
Locations (1):
- ViRx Inc, San Francisco, California, United States

REFERENCES:
- [Background] Gordon M, Guralnik M, Kaneko Y, Mimura T, Baker M, Lang W. A phase I study of curdlan sulfate--an HIV inhibitor. Tolerance, pharmacokinetics and effects on coagulation and on CD4 lymphocytes. J Med. 1994;25(3-4):163-80. PMID 7996061